CLINICAL TRIAL: NCT06594744
Title: A Randomized Controlled Trial of Endoscopic Variceal Ligation Versus Carvedilol for the Prevention of First Esophageal Variceal Bleeding in Patients With Hepatocellular Carcinoma
Brief Title: Endoscopic Variceal Ligation vs Carvedilol for the Prevention of First Esophageal Variceal Bleeding in Patients With HCC
Acronym: P-HCC-CVL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02-016B
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma (HCC); Esophageal Varices
Keywords: Endoscopic variceal ligation; Hepatocellular carcinoma; Nonselective beta-blocker; Portal hypertension
MeSH Terms: conditions — Carcinoma, Hepatocellular; Esophageal and Gastric Varices; Hypertension, Portal | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: EVL group:
  EVL will be performed and repeated every 3 to 4 weeks until the EVs are eradicated. Following this, patients will undergo regular upper gastrointestinal endoscopic surveillance, initially every three months for a total of two sessions, then every six months for a total of two sessions, and subsequently annually. If EVs are found to recur during surveillance, additional EVL will be performed every 3 to 4 weeks until the varices are again eradicated endoscopically.
  Carvedilol group:
  The initial dosage of carvedilol is set at 6.25 mg daily. In the absence of hypotension (systolic blood pressure < 90 mmHg), bradycardia (resting heart rate < 55 beats per minute), or other adverse effects, hospitalized patients may have their dosage increased to 12.5 mg daily after 3 days, while outpatient patients may increase their dosage to 12.5 mg daily after 7 days. This dosage represents the target dose for the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic variceal ligation (Active Comparator): EVL will be performed and repeated every 3 to 4 weeks until the EVs are eradicated. Following this, patients will undergo regular upper gastrointestinal endoscopic surveillance, initially every three months for a total of two sessions, then every six months for a total of two sessions, and subsequently annually. If EVs are found to recur during surveillance, additional EVL will be performed every 3 to 4 weeks until the varices are again eradicated endoscopically.
  Interventions: Procedure: Endoscopic variceal ligation
- Carvedilol (Placebo Comparator): The initial dosage of carvedilol is set at 6.25 mg daily. In the absence of hypotension (systolic blood pressure < 90 mmHg), bradycardia (resting heart rate < 55 beats per minute), or other adverse effects, hospitalized patients may have their dosage increased to 12.5 mg daily after 3 days, while outpatient patients may increase their dosage to 12.5 mg daily after 7 days. This dosage represents the target dose for the trial.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Procedure: Endoscopic variceal ligation — EVL will be performed and repeated every 3 to 4 weeks until the EVs are eradicated. Following this, patients will undergo regular upper gastrointestinal endoscopic surveillance, initially every three months for a total of two sessions, then every six months for a total of two sessions, and subsequently annually. If EVs are found to recur during surveillance, additional EVL will be performed every 3 to 4 weeks until the varices are again eradicated endoscopically.
  Arms: Endoscopic variceal ligation
Drug: Carvedilol — The initial dosage of carvedilol is set at 6.25 mg daily. In the absence of hypotension (systolic blood pressure < 90 mmHg), bradycardia (resting heart rate < 55 beats per minute), or other adverse effects, hospitalized patients may have their dosage increased to 12.5 mg daily after 3 days, while outpatient patients may increase their dosage to 12.5 mg daily after 7 days. This dosage represents the target dose for the trial.
  Arms: Carvedilol

SUMMARY:
The goal of this clinical trial is to evaluate whether endoscopic variceal ligation (EVL) or carvedilol is more effective at preventing the first esophageal variceal bleeding (EVB) in patients with hepatocellular carcinoma (HCC). It will also learn about the safety of EVL and carvedilol in patients with HCC. The main questions it aims to answer are:

Whether EVL or carvedilol is more effective at preventing initial EVB in patients with HCC with high-risk EVs.

What medical problems do participants have when undergoing EVL or taking carvedilol? Researchers will compare the efficacy and safety of EVL to carvedilol for the prevention of first EVB in patients with HCC.

Participants will:

Undergo EVL every 3-4 weeks until variceal eradication and then receive regular endoscopic follow-up according to the protocol, or Take carvedilol every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable).

Visit the clinic once every 2-3 months for checkups and tests. Keep a diary of their vital signs (SBP, DBP, and HR) as well as symptoms.

DETAILED DESCRIPTION:
Gastro-esophageal variceal bleeding is a major complication of portal hypertension (PHT) and carries a high rate of rebleeding and mortality. Hepatocellular carcinoma (HCC), a special subgroup of PHT, is the sixth most commonly diagnosed cancer and the third leading cause of cancer death worldwide. The presence of esophageal varices (EVs) in more than half of patients with HCC is associated with poor survival. Furthermore, without primary prevention strategies, nearly half of these HCC patients experience esophageal variceal bleeding (EVB). The prognosis of HCC patients with EVB is extremely poor, with a rebleeding rate of 50% and a six-week mortality rate of 26-48%, both of which are higher than those of non-HCC patients.

However, there is still a lack of evidence on how to prevent first EVB in patients with HCC with high-risk EVs. AASLD practice guidance recommends prevention of EVB and hepatic decompensation in patients with HCC should follow the same principles as those for patients without HCC, that is, nonselective beta-blocker (NSBB) therapy is recommended in patients with HCC with clinically significant portal hypertension (CSPH). Endoscopic variceal ligation (EVL) is recommended for compensated patients with high-risk EVs who have contraindications to NSBBs. However, this recommendation lacks randomized controlled trial (RCT) to support it. Our recently published RCT showed that EVL is superior to propranolol (PPL) in the primary prevention of EVB in patients with HCC with high-risk EVs. In the subgroup analysis, EVL reduces EVB and improves OS in patients with BCLC stage A/B but not in those with BCLC stage C/D.

Carvedilol, an NSBB that additionally exerts intrinsic anti-alpha-1-adrenergic activity, has been shown to reduce hepatic venous pressure gradient more than propranolol and is currently the first-line treatment for primary prophylaxis in patients with CSPH. Nevertheless, the superiority of EVL versus carvedilol as a primary prevention strategy in patients with HCC with high-risk EVs is still unknown. In this project, we will initiate an open-label RCT aiming at comparing the efficacy of EVL and carvedilol in the primary prevention of EVB in patients with HCC with high-risk EVs. We will also explore if there is any difference between the two groups in terms of other upper gastrointestinal bleeding, nonbleeding liver decompensation (such as new onset/worsening ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, and hepatorenal syndrome), overall survival, adverse events, tolerability and safety. We will also compare the efficacy of EVL and carvedilol in the primary prevention of EVB in patients with HCC at different BCLC stage.

ELIGIBILITY:
Inclusion Criteria:

- Patients with HCC and high-risk EVs, confirmed through imaging and clinical data (classified as F2 or F3 EVs according to Beppu et al. classification)

Exclusion Criteria:

* Age less than 20 years or greater than 90 years.
* History of esophageal variceal bleeding.
* Previous treatment for EVs, including EVL, endoscopic sclerotherapy, transjugular intrahepatic portosystemic shunt (TIPS), or surgical interventions.
* Use of non-selective β-blockers within two weeks prior to enrollment.
* Contraindications for non-selective β-blockers, including severe atrioventricular block, chronic obstructive pulmonary disease (COPD), asthma, poorly controlled diabetes, and severe peripheral artery disease.
* Presence of other end-stage organ diseases, including terminal cancers other than HCC, heart failure, and renal failure.
* Pregnant women.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Esophageal variceal bleeding | 3 years
  The cumulative incidence of esophageal variceal bleeding

SECONDARY OUTCOMES:
Other upper gastrointestinal bleeding | 3 years
  The cumulative incidence of other upper gastrointestinal bleeding
First/further nonbleeding liver decompensation | 3 years
  Events that defined first/further nonbleeding liver decompensation were based on the Baveno VII consensus
Overall survival | 3 years
Adverse events | 3 years

OTHER OUTCOMES:
Primary and secondary outcomes categorized by BCLC staging in the subgroup analysis | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan DE, Ripoll C, Thiele M, Fortune BE, Simonetto DA, Garcia-Tsao G, Bosch J. AASLD Practice Guidance on risk stratification and management of portal hypertension and varices in cirrhosis. Hepatology. 2024 May 1;79(5):1180-1211. doi: 10.1097/HEP.0000000000000647. Epub 2023 Oct 23. No abstract available. PMID 37870298
- [Background] Llovet JM, Bru C, Bruix J. Prognosis of hepatocellular carcinoma: the BCLC staging classification. Semin Liver Dis. 1999;19(3):329-38. doi: 10.1055/s-2007-1007122. PMID 10518312
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Sarin SK, Lahoti D, Saxena SP, Murthy NS, Makwana UK. Prevalence, classification and natural history of gastric varices: a long-term follow-up study in 568 portal hypertension patients. Hepatology. 1992 Dec;16(6):1343-9. doi: 10.1002/hep.1840160607. PMID 1446890
- [Background] Beppu K, Inokuchi K, Koyanagi N, Nakayama S, Sakata H, Kitano S, Kobayashi M. Prediction of variceal hemorrhage by esophageal endoscopy. Gastrointest Endosc. 1981 Nov;27(4):213-8. doi: 10.1016/s0016-5107(81)73224-3. PMID 6975734
- [Background] Serper M, Kaplan DE, Taddei TH, Tapper EB, Cohen JB, Mahmud N. Nonselective beta blockers, hepatic decompensation, and mortality in cirrhosis: A national cohort study. Hepatology. 2023 Feb 1;77(2):489-500. doi: 10.1002/hep.32737. Epub 2022 Oct 17. PMID 35984731
- [Background] Kalambokis GN, Christaki M, Tsiakas I, Despotis G, Fillipas-Ntekouan S, Fotopoulos A, Tsiouris S, Xourgia X, Lakkas L, Pappas K, Michalis LK, Sergianiti F, Baltayiannis G, Christodoulou D, Koustousi C, Aggelis N, Milionis H. Conversion of Propranolol to Carvedilol Improves Renal Perfusion and Outcome in Patients With Cirrhosis and Ascites. J Clin Gastroenterol. 2021 Sep 1;55(8):721-729. doi: 10.1097/MCG.0000000000001431. PMID 32991355
- [Background] Totzeck M, Mincu RI, Rassaf T. Cardiovascular Adverse Events in Patients With Cancer Treated With Bevacizumab: A Meta-Analysis of More Than 20 000 Patients. J Am Heart Assoc. 2017 Aug 10;6(8):e006278. doi: 10.1161/JAHA.117.006278. PMID 28862931
- [Background] Abou-Alfa GK, Lau G, Kudo M, Chan SL, Kelley RK, Furuse J, Sukeepaisarnjaroen W, Kang YK, Van Dao T, De Toni EN, Rimassa L, Breder V, Vasilyev A, Heurgue A, Tam VC, Mody K, Thungappa SC, Ostapenko Y, Yau T, Azevedo S, Varela M, Cheng AL, Qin S, Galle PR, Ali S, Marcovitz M, Makowsky M, He P, Kurland JF, Negro A, Sangro B. Tremelimumab plus Durvalumab in Unresectable Hepatocellular Carcinoma. NEJM Evid. 2022 Aug;1(8):EVIDoa2100070. doi: 10.1056/EVIDoa2100070. Epub 2022 Jun 6. PMID 38319892
- [Background] Cheng AL, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Lim HY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Ma N, Nicholas A, Wang Y, Li L, Zhu AX, Finn RS. Updated efficacy and safety data from IMbrave150: Atezolizumab plus bevacizumab vs. sorafenib for unresectable hepatocellular carcinoma. J Hepatol. 2022 Apr;76(4):862-873. doi: 10.1016/j.jhep.2021.11.030. Epub 2021 Dec 11. PMID 34902530
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Allaire M, Thabut D. Portal hypertension and variceal bleeding in patients with liver cancer: Evidence gaps for prevention and management. Hepatology. 2024 Jan 1;79(1):213-223. doi: 10.1097/HEP.0000000000000291. Epub 2023 Jan 13. PMID 36631021
- [Background] Thabut D, Kudo M. Treatment of portal hypertension in patients with HCC in the era of Baveno VII. J Hepatol. 2023 Mar;78(3):658-662. doi: 10.1016/j.jhep.2022.11.019. Epub 2022 Nov 30. PMID 36460163
- [Background] Shah HA, Azam Z, Rauf J, Abid S, Hamid S, Jafri W, Khalid A, Ismail FW, Parkash O, Subhan A, Munir SM. Carvedilol vs. esophageal variceal band ligation in the primary prophylaxis of variceal hemorrhage: a multicentre randomized controlled trial. J Hepatol. 2014 Apr;60(4):757-64. doi: 10.1016/j.jhep.2013.11.019. Epub 2013 Nov 28. PMID 24291366
- [Background] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Background] Tripathi D, Ferguson JW, Kochar N, Leithead JA, Therapondos G, McAvoy NC, Stanley AJ, Forrest EH, Hislop WS, Mills PR, Hayes PC. Randomized controlled trial of carvedilol versus variceal band ligation for the prevention of the first variceal bleed. Hepatology. 2009 Sep;50(3):825-33. doi: 10.1002/hep.23045. PMID 19610055
- [Background] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2019 Apr 20;393(10181):1597-1608. doi: 10.1016/S0140-6736(18)31875-0. Epub 2019 Mar 22. PMID 30910320
- [Background] Villanueva C, Torres F, Sarin SK, Shah HA, Tripathi D, Brujats A, Rodrigues SG, Bhardwaj A, Azam Z, Hayes PC, Jindal A, Abid S, Alvarado E, Bosch J; Carvedilol-IPD-MA-group and the Baveno Cooperation: an EASL Consortium. Carvedilol reduces the risk of decompensation and mortality in patients with compensated cirrhosis in a competing-risk meta-analysis. J Hepatol. 2022 Oct;77(4):1014-1025. doi: 10.1016/j.jhep.2022.05.021. Epub 2022 May 31. PMID 35661713
- [Background] Jachs M, Hartl L, Simbrunner B, Bauer D, Paternostro R, Balcar L, Hofer B, Pfisterer N, Schwarz M, Scheiner B, Stattermayer AF, Pinter M, Trauner M, Mandorfer M, Reiberger T. Carvedilol Achieves Higher Hemodynamic Response and Lower Rebleeding Rates Than Propranolol in Secondary Prophylaxis. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2318-2326.e7. doi: 10.1016/j.cgh.2022.06.007. Epub 2022 Jul 14. PMID 35842118
- [Background] Jutabha R, Jensen DM, Martin P, Savides T, Han SH, Gornbein J. Randomized study comparing banding and propranolol to prevent initial variceal hemorrhage in cirrhotics with high-risk esophageal varices. Gastroenterology. 2005 Apr;128(4):870-81. doi: 10.1053/j.gastro.2005.01.047. PMID 15825071
- [Background] Schepke M, Kleber G, Nurnberg D, Willert J, Koch L, Veltzke-Schlieker W, Hellerbrand C, Kuth J, Schanz S, Kahl S, Fleig WE, Sauerbruch T; German Study Group for the Primary Prophylaxis of Variceal Bleeding. Ligation versus propranolol for the primary prophylaxis of variceal bleeding in cirrhosis. Hepatology. 2004 Jul;40(1):65-72. doi: 10.1002/hep.20284. PMID 15239087
- [Background] Lui HF, Stanley AJ, Forrest EH, Jalan R, Hislop WS, Mills PR, Finlayson ND, Macgilchrist AJ, Hayes PC. Primary prophylaxis of variceal hemorrhage: a randomized controlled trial comparing band ligation, propranolol, and isosorbide mononitrate. Gastroenterology. 2002 Sep;123(3):735-44. doi: 10.1053/gast.2002.35385. PMID 12198700
- [Background] Sarin SK, Lamba GS, Kumar M, Misra A, Murthy NS. Comparison of endoscopic ligation and propranolol for the primary prevention of variceal bleeding. N Engl J Med. 1999 Apr 1;340(13):988-93. doi: 10.1056/NEJM199904013401302. PMID 10099140
- [Background] Lim J, Kim HI, Kim E, Kim J, An J, Chang S, Kim SO, Lee HC, Lee YS, Shim JH. Variceal bleeding is aggravated by portal venous invasion of hepatocellular carcinoma: a matched nested case-control study. BMC Cancer. 2021 Jan 5;21(1):11. doi: 10.1186/s12885-020-07708-1. PMID 33402105
- [Background] Sidali S, Nault JC. Portal hypertension and hepatocellular carcinoma: Navigating uncharted waters. United European Gastroenterol J. 2022 Feb;10(1):8-9. doi: 10.1002/ueg2.12193. Epub 2022 Jan 8. No abstract available. PMID 34997990
- [Background] Allaire M, Rudler M, Thabut D. Portal hypertension and hepatocellular carcinoma: Des liaisons dangereuses.... Liver Int. 2021 Aug;41(8):1734-1743. doi: 10.1111/liv.14977. Epub 2021 Jun 28. PMID 34051060
- [Background] Ripoll C, Groszmann RJ, Garcia-Tsao G, Bosch J, Grace N, Burroughs A, Planas R, Escorsell A, Garcia-Pagan JC, Makuch R, Patch D, Matloff DS; Portal Hypertension Collaborative Group. Hepatic venous pressure gradient predicts development of hepatocellular carcinoma independently of severity of cirrhosis. J Hepatol. 2009 May;50(5):923-8. doi: 10.1016/j.jhep.2009.01.014. Epub 2009 Mar 5. PMID 19303163
- [Background] Kadouchi K, Higuchi K, Shiba M, Okazaki H, Yamamori K, Sasaki E, Tominaga K, Watanabe T, Fujiwara Y, Oshitani N, Arakawa T. What are the risk factors for aggravation of esophageal varices in patients with hepatocellular carcinoma? J Gastroenterol Hepatol. 2007 Feb;22(2):240-6. doi: 10.1111/j.1440-1746.2006.04418.x. PMID 17295878
- [Background] Yang TC, Chen WC, Hou MC, Chen PH, Lee PC, Chang CY, Lu HS, Chen YJ, Hsu SJ, Huang HC, Luo JC, Huang YH, Lee FY. Endoscopic variceal ligation versus propranolol for the primary prevention of oesophageal variceal bleeding in patients with hepatocellular carcinoma: an open-label, two-centre, randomised controlled trial. Gut. 2024 Mar 7;73(4):682-690. doi: 10.1136/gutjnl-2023-330419. PMID 38123994
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Kim JH, Sinn DH, Kim K, Kang W, Gwak GY, Paik YH, Choi MS, Lee JH, Koh KC, Paik SW. Primary Prophylaxis for Variceal Bleeding and the Improved Survival of Patients with Newly Diagnosed Hepatocellular Carcinoma. Dig Dis Sci. 2016 Nov;61(11):3354-3362. doi: 10.1007/s10620-016-4255-6. Epub 2016 Jul 19. PMID 27435325
- [Background] Chen WC, Hou MC, Lin HC, Lee FY, Yeh YY, Chang FY, Lee SD. Feasibility and potential benefit of maintenance endoscopic variceal ligation in patients with unresectable hepatocellular carcinoma and acute esophageal variceal hemorrhage: a controlled trial. Gastrointest Endosc. 2001 Jul;54(1):18-23. doi: 10.1067/mge.2001.115731. PMID 11427836
- [Background] Akahoshi T, Tomikawa M, Tsutsumi N, Hashizume M, Maehara Y. Merits of prophylactic sclerotherapy for esophageal varices concomitant unresectable hepatocellular carcinoma: prospective randomized study. Dig Endosc. 2014 Mar;26(2):172-7. doi: 10.1111/den.12119. Epub 2013 May 8. PMID 23650913
- [Background] Iwakiri R, Koyama T, Hirano M, Uchida Y, Ishibashi S, Kuwahara A, Matsunaga K, Sakata H, Fujimoto K. Endoscopic injection sclerotherapy for esophageal varices prolonged survival of patients with hepatocellular carcinoma complicating liver cirrhosis. Gastrointest Endosc. 2000 May;51(5):569-72. doi: 10.1016/s0016-5107(00)70291-4. PMID 10805843
- [Background] Miyoshi H, Matsumoto A, Oka M, Sugi K, Yoshimura K, Hongou Y, Katsu K. Efficacy of prophylactic sclerotherapy in patients with hepatocellular carcinoma and varices negative for the red color sign. Gastrointest Endosc. 1997 Jun;45(6):498-502. doi: 10.1016/s0016-5107(97)70180-9. PMID 9199908
- [Background] Bucci L, Garuti F, Camelli V, Lenzi B, Farinati F, Giannini EG, Ciccarese F, Piscaglia F, Rapaccini GL, Di Marco M, Caturelli E, Zoli M, Borzio F, Sacco R, Maida M, Felder M, Morisco F, Gasbarrini A, Gemini S, Foschi FG, Missale G, Masotto A, Affronti A, Bernardi M, Trevisani F; Italian Liver Cancer (ITA.LI.CA) Group; Italian Liver Cancer ITA LI CA Group. Comparison between alcohol- and hepatitis C virus-related hepatocellular carcinoma: clinical presentation, treatment and outcome. Aliment Pharmacol Ther. 2016 Feb;43(3):385-99. doi: 10.1111/apt.13485. Epub 2015 Dec 14. PMID 26662476
- [Background] Giannini EG, Risso D, Testa R, Trevisani F, Di Nolfo MA, Del Poggio P, Benvegnu L, Ludovico Rapaccini G, Farinati F, Zoli M, Borzio F, Caturelli E; Italian Liver Cancer (ITA.LI.CA.) Group. Prevalence and prognostic significance of the presence of esophageal varices in patients with hepatocellular carcinoma. Clin Gastroenterol Hepatol. 2006 Nov;4(11):1378-84. doi: 10.1016/j.cgh.2006.08.011. Epub 2006 Oct 23. PMID 17059899
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Lee YR, Park SY, Tak WY. Treatment Outcomes and Prognostic Factors of Acute Variceal Bleeding in Patients with Hepatocellular Carcinoma. Gut Liver. 2020 Jul 15;14(4):500-508. doi: 10.5009/gnl19155. PMID 31816673
- [Background] Garcia-Tsao G, Lim JK; Members of Veterans Affairs Hepatitis C Resource Center Program. Management and treatment of patients with cirrhosis and portal hypertension: recommendations from the Department of Veterans Affairs Hepatitis C Resource Center Program and the National Hepatitis C Program. Am J Gastroenterol. 2009 Jul;104(7):1802-29. doi: 10.1038/ajg.2009.191. Epub 2009 May 19. PMID 19455106
- [Background] El-Serag HB, Everhart JE. Improved survival after variceal hemorrhage over an 11-year period in the Department of Veterans Affairs. Am J Gastroenterol. 2000 Dec;95(12):3566-73. doi: 10.1111/j.1572-0241.2000.03376.x. PMID 11151893
- [Background] Sanyal AJ, Bosch J, Blei A, Arroyo V. Portal hypertension and its complications. Gastroenterology. 2008 May;134(6):1715-28. doi: 10.1053/j.gastro.2008.03.007. No abstract available. PMID 18471549